CLINICAL TRIAL: NCT05843123
Title: Comparison of Carbon Dioxide Control During Pressure Controlled (PC) Versus Pressure Regulated Volume Control (PRVC) Ventilation in Children (CoCO2): a Digital, Randomized Controlled Trial
Brief Title: Comparison of Gas Exchange Between Two Invasive Mechanical Ventilation Modes in Children
Acronym: CoCO2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CoCO2
Record Dates: First submitted 2023-01-24; First posted 2023-05-06 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Respiratory Failure
Keywords: Pediatrics; Child; Infant; Mechanical ventilation; Pressure control; Pressure regulated volume control; Randomized controlled trial
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: This is a single center, open labelled, randomized controlled trial with one to one allocation to two invasive mechanical ventilation modes used in clinical care as intervention arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pressure control (PC) (Active Comparator): In PC physicians set the inspiratory pressure and time, the respiratory rate and the PEEP while the ventilator measures tidal volume and the actual respiratory rate
  Interventions: Other: Respiratory support b
- Pressure regulated volume control (PRVC) (Active Comparator): In PRVC physicians set a target tidal volume and the respiratory rate. An algorithm delivers pressure using a decelerating flow pattern to reach the target tidal volume based on the lung compliance measured during previous breaths.
  Interventions: Other: Respiratory support a

INTERVENTIONS:
Other: Respiratory support a — Invasive mechanical ventilation mode
  Other Names: "Target Vent" is the brand name of the PRVC ventilation mode in the Bellavista ventilator
  Arms: Pressure regulated volume control (PRVC)
Other: Respiratory support b — Invasive mechanical ventilation mode
  Arms: Pressure control (PC)

SUMMARY:
This study assesses the feasibility of digital data collection for a randomized controlled trial in a quaternary pediatric intensive care unit and the effect of two commonly used mechanical ventilation modes on gas exchange (CO2) in children over 2 days after randomization.

This is a single-center, open-labelled, randomized controlled trial with two parallel 1:1 treatment arms: pressure controlled (PC) vs pressure-regulated volume controlled (PRVC) mechanical ventilation modes.

Use to routine digital data is essential to enable health learning systems and to provide rapid clinical trials readiness, as the pandemic has demonstrated. Despite availability of data to perform digital trials in PICU settings, these are yet scarcely done.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent provided by the participant or the participant's parents or legal guardians. In case of an emergency situation, a physician who is independent of the research project must be consulted prior to inclusion in order to safeguard the interests of the test subject.
* Admission to PICU at the University Children's Hospital Zurich
* Need for mechanical ventilation for >60 min during PICU hospitalization. Need for mechanical ventilation will be based on clinical decision of the treating physician.
* Need for an arterial line during PICU hospitalization. Need for an arterial line will be based on clinical decision of the treating physician.
* Age <18 years
* Weight >2 Kg

Exclusion Criteria:

* Substantial air leaks around the endotracheal tube (>30%)
* Cyanotic shunt lesions
* Intracranial hypertension (i.e. traumatic brain injury or patients admitted after neurosurgery)
* Pulmonary hypertension under treatment (i.e sildenafil or inhaled nitric oxide)
* Time from start of invasive mechanical ventilation until time of screening is > 24 hours
* Previous enrolment in the study in the past 30 days
* Inability of the parents or legal guardians to understand the study due to linguistic or cognitive reasons

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 59 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
Adherence to the allocated ventilation mode among randomized/enrolled participants | From time of randomization until 48 hours, extubation, discharge or death, whichever comes first (assessed up to 48 hours)
  Main feasibility outcome
Proportion of time spent within the target range of carbon dioxide (normocarbia, defined as carbon dioxide ≥ 35 mmHg or 4.5 kPa and ≤ 45 mmHg or 6 kPa) measured using end-tidal carbon dioxide recorded every minute by the ventilation device | From time of randomization until 48 hours, extubation, discharge or death, whichever comes first (assessed up to 48 hours)
  Main physiological outcome

SECONDARY OUTCOMES:
Number of patients who were screened, were missed, gave consent and were randomized/enrolled per month | From date of recruitment start until date of recruitment end (assessed when n=60, anticipated through 6 months of recruitment period)
  Secondary feasibility outcome 1
Reasons for protocol violations | From time of randomization until 48 hours, extubation, discharge or death, whichever comes first (assessed up to 48 hours since randomization)
  Other feasibility outcome 2a
Time from randomization to protocol violation | From time of randomization until time of protocol violation (assessed up to 48 hours)
  Other feasibility outcome 2b
Proportion of enrolled participants with complete primary and secondary outcome data extracted from the electronic patient records | From date of recruitment start until date of study end (assessed when n=60 and data has been extracted for all participants, anticipated through 8 months)
  Other feasibility outcome 3
Time from ventilation start until screening | From time of ventilation start until time of screening (assessed up to 48 hours)
  Other feasibility outcome 4a
Time from ventilation start until randomization | From time of ventilation start until time of randomization (assessed up to 48 hours)
  Other feasibility outcome 4b
Time from consent until randomization | From time of consent signed until time of randomization (assessed up to 48 hours)
  Other feasibility outcome 5
Time weighted average of hypocarbia (carbon dioxide < 35 mmHg or 4.5 kPa), measured using continuous end-tidal carbon dioxide | From time of randomization until 48 hours, extubation, discharge or death, whichever comes first (assessed up to 48 hours)
  Secondary physiological outcome 1a
Time weighted average of hypocarbia (carbon dioxide < 35 mmHg or 4.5 kPa) measured using intermittent arterial blood measurements | From time of randomization until 48 hours, extubation, discharge or death, whichever comes first (assessed up to 48 hours)
  Other physiological outcome 1b
Time weighted average of hypocarbia (carbon dioxide < 35 mmHg or 4.5 kPa) measured using continuous transcutaneous carbon dioxide measurements calibrated with results of arterial blood gas analysis | From time of randomization until 48 hours, extubation, discharge or death, whichever comes first (assessed up to 48 hours)
  Other physiological outcome 1c
Time weighted average of hypercarbia (carbon dioxide > 45 mmHg or 6 kPa) measured using continuous end-tidal carbon dioxide | From time of randomization until 48 hours, extubation, discharge or death, whichever comes first (assessed up to 48 hours)
  Other physiological outcome 2a
Time weighted average of hypercarbia (carbon dioxide >45 mmHg or 6 kPa) measured using intermittent arterial blood measurements | From time of randomization until 48 hours, extubation, discharge or death, whichever comes first (assessed up to 48 hours)
  Other physiological outcome 2b
Time weighted average of hypercarbia (carbon dioxide > 45 mmHg or 6 kPa) measured using continuous transcutaneous carbon dioxide measurements calibrated with results of arterial blood gas analysis | From time of randomization until 48 hours, extubation, discharge or death, whichever comes first (assessed up to 48 hours)
  Other physiological outcome 2c
Time weighted average of hypo- and hypercarbia (i.e. outside normocarbia, carbon dioxide < 35 mmHg or 4.5 kPa; or carbon dioxide >45 mmHg or 6 kPa) measured using continuous end-tidal carbon dioxide | From time of randomization until 48 hours, extubation, discharge or death, whichever comes first (assessed up to 48 hours)
  Other physiological outcome 3a
Time weighted average of hypo- and hypercarbia (i.e. outside normocarbia, carbon dioxide < 35 mmHg or 4.5 kPa; or carbon dioxide >45 mmHg or 6 kPa) measured using intermittent arterial blood measurements | From time of randomization until 48 hours, extubation, discharge or death, whichever comes first (assessed up to 48 hours)
  Other physiological outcome 3b
Time weighted average of hypo- and hypercarbia (i.e. carbon dioxide < 35 mmHg or 4.5 kPa; or >45 mmHg or 6 kPa) measured using continuous transcutaneous carbon dioxide measurements calibrated with results of arterial blood gas analysis | From time of randomization until 48 hours, extubation, discharge or death, whichever comes first (assessed up to 48 hours)
  Other physiological outcome 3c

OTHER OUTCOMES:
Oxygenation index measured using peripheral oxygen saturation index | From time of randomization until 48 hours, extubation, discharge or death, whichever comes first (assessed up to 48 hours)
  Other physiological outcome 4a (Peripheral oxygen saturation index = MAP * FiO2 *100 / SpO2; where MAP is mean airway pressure, FiO2 is fraction of inspired oxygen, SpO2 is peripheral oxygen saturation)
Oxygenation index measured using arterial oxygenation index | From time of randomization until 48 hours, extubation, discharge or death, whichever comes first (assessed up to 48 hours)
  Other physiological outcome 4b (Arterial oxygenation index = MAP * FiO2 *100 / PaO2 ; where MAP is mean airway pressure, FiO2 is fraction of inspired oxygen, PaO2 is partial pressure of oxygen in arterial blood)

CONTACTS AND LOCATIONS:
Overall Officials: Rebeca Mozun, MD PhD, Principal Investigator — University Children's Hospital, Zurich
Locations (1):
- University Children's Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
The research team will have access to the dataset of this study. Anonymized data could be available upon reasonable request after approval from the research committee and sponsoring institution.

REFERENCES:
- [Derived] Mozun R, Chopard D, Zapf F, Baumann P, Brotschi B, Adam A, Jaeggi V, Bangerter B, Gibbons KS, Burren J, Schlapbach LJ. Comparison of carbon dioxide control during pressure controlled versus pressure-regulated volume controlled ventilation in children (CoCO2): protocol for a pilot digital randomised controlled trial in a quaternary paediatric intensive care unit. BMJ Open. 2025 Jan 11;15(1):e087043. doi: 10.1136/bmjopen-2024-087043. PMID 39800404